CLINICAL TRIAL: NCT03622086
Title: Foundations of Fitness: A Clinic-Community Partnership to Address Pediatric Obesity
Brief Title: Foundations of Fitness Program Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Auden McClure, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D18143
Record Dates: First submitted 2018-07-18; First posted 2018-08-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Pediatric Obesity; Health Behavior; Body Mass Index; Self Esteem
MeSH Terms: conditions — Pediatric Obesity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-10 years old (Experimental): Children-caregiver pairs will participate in a 24-week pilot that includes 2 phases, 12 weeks of usual care, followed by 12 weeks of Foundations of Fitness Program.
  Interventions: Other: Foundations of Fitness Program
- 11-13 years old (Experimental): Children-caregiver pairs will participate in a 24-week pilot that includes 2 phases, 12 weeks of usual care, followed by 12 weeks of Foundations of Fitness Program.
  Interventions: Other: Foundations of Fitness Program

INTERVENTIONS:
Other: Foundations of Fitness Program — The Foundations of Fitness Program is a 12 week, bi-weekly community intensive lifestyle program which focuses on healthy diet, daily physical activity, self-esteem and support for individual and family behavior change, components supported by USPSTF evidence review. Class sessions, which involve both parent/caregiver and child will include structured fitness activities, hands on nutrition, cooking, shopping and meal planning and facilitated discussions about goal setting, self-monitoring, stimulus control and healthy homes and families. Content will be offered in a context that supports self-esteem and behavior change. The program was developed by the Carter Community Building Association (CCBA) in collaboration with the Dartmouth-Hitchcock Weight & Wellness Center research core.

SUMMARY:
Approximately 17% of US children have obesity resulting in significant childhood co-morbidities and increased lifetime risk of adult obesity, diabetes, cardiovascular disease and cancer. Guidelines recommend intensive lifestyle programs as first-line treatment, yet few pediatric practices are equipped to provide this. Clinical-community partnerships are well-positioned to address this care gap. This proposal aims to assess whether a community-delivered lifestyle program offered in adjunct to primary care obesity management is feasible, acceptable, effective, and easily implemented in a rural care setting. In this study, approximately 40 children aged 7-13 years old and their caregiver pairs will be recruited from a primary care pediatric clinic. Child-adult dyads will participate in a 24-week program that includes 2 phases, a 12-week usual care phase and a 12-week intervention phase. The intervention phase will include bi-weekly meetings of a community intensive lifestyle program which focuses on healthy diet, daily physical activity, self-esteem and support for individual and family behavior change. A mixed-methods approach using qualitative interviews and study questionnaires, combined with objective measures of adiposity and fitness will assess study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-13 years;
* BMI% ≥85th%;
* Regional pediatric medical home patient;
* English speaking child and parent/caregiver;

Exclusion Criteria:

* Physical or developmental limitation to participation as determined by referring provider

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Program Feasibility based on program attendance and completion of assessments to determine if children are willing and interested in to attending a fitness program. | 24 weeks
  Programmatic feasibility will be defined as delivery of 100% of the sessions with 80% of children attending ≥75% of sessions and 80% completing pre- and post-assessments.
Program Acceptability based on interviews evaluating the appropriateness of the pilot and assessing strengths/weaknesses. | 24 weeks
  Program acceptability will be assessed through semi-structured participant interviews ensuring the appropriateness of the pilot and assessing strengths/weaknesses.
Program Eligibility rate | 24 weeks
  Calculated using the following formula: [# screen positive / # screened for inclusion].
Program Enrollment rate | 24 weeks
  Calculated using the following formula: [# enrolled / (# screen positive & eligible)]. We will assess reasons for dropout/non-adherence.
Program Completion rate | 24 weeks
  Calculated using the following formula: (# completing all sessions / # enrolled).
Assessment Completion rate | 24 weeks
  Calculated using the following formula: (# completing all assessments / # enrolled).
Participant Satisfaction Survey | 24 weeks
  A 12 item survey at program conclusion will assess patient satisfaction with program elements (overall, class sessions, staff, assessments) using Likert scales (1-5 point scale - very dissatisfied=1 to very satisfied=5).

SECONDARY OUTCOMES:
Body Mass Index Percentile | 48 weeks
  Height (cm) and Weight (kg) will be used to calculate body mass index (kg/m^2) and then BMI percentile (%) using Center for Disease Control 2000 standards.
Strength Assessment | 24 weeks
  Assessed through 5 exercises including: leg extension, leg curl, lap pull down, shoulder press, chest press. Units for all are number of repetitions per minute at a fixed mass (lbs).
Health Habits Survey | 24 weeks
  The Weight & Wellness Center Health Habits Survey assesses diet, activity, media and sleep behaviors through 46 individual survey questions with variable response categories (for example, overall physical activity is assessed using a 0-5 point Likert scale with higher score related to better physical activity level: " Overall my physical activity level is": Poor=0 - Excellent=5)
Subjective Health and Quality of Life Score | 24 weeks
  The Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Health 7 survey (child and parent proxy) is a 7-question survey (Score 7-35) capturing physical, mental, and social aspects of quality of life using Likert scales (1-5 point scale: poor/never=1 to excellent/always=5). Higher score indicates more positive perceptions of overall health.
Sense of Belonging in Fitness Program Score | 24 weeks
  The Anderson-Butcher and Conroy Sense of Belonging survey is a 5-item questionnaire measuring sense of belonging experienced by children participating in a Fitness Program using Likert scale (1-4 point scale: NO!=1, no=2, yes=3, and YES!=4). Total Score Range 5-20: A higher score indicates a greater sense of belonging.
Self Esteem Score | 24 weeks
  The Rosenberg Self-Esteem survey is a 10-item questionnaire measuring self-esteem of children participating in a Fitness Program using Likert scale (0-3 point scale: Strongly disagree=0 to Strongly agree=3). Total Score Range 0-30: Higher scores indicate greater self-esteem.
Physical Activity Score | 24 weeks
  The Patient Reported Outcomes Measurement Information Systems (PROMIS) is a short form 4-question survey (Score 4-20) assessing physical activity over the past seven days using Likert scales (1-5 point scale: No days=1, 1 day=2, 2-3 days=3, 4-5 days=4, and 6-7 days=5). Higher score indicates higher levels of physical activity.
Cardio-capacity | 24 weeks
  Distance (m) on treadmill at 65% of max heart rate.
Heart Rate | 24 weeks
  Resting and recovery heart rate (BPM) measured before and after treadmill test.
Blood Pressure | 24 weeks
  Resting and recovery systolic and diastolic Blood pressure (mmHg) measured before and after treadmill test.
Waist Circumference | 24 weeks
  Waist circumference will be measured (cm)
Perceived Athletic Competence Score | 24 weeks
  The Harter Self-Perception Profile for Children is a short form 6-question survey (score 1-4) assessing athletic competence using a two-choice format with option then of checking "Sort of True for Me" or "Really True for Me" (A score of 1 indicates lowest and a score of 4 highest level of perceived athletic competence).

OTHER OUTCOMES:
Staff program adoption | 24 weeks
  Staff program adoption will be assessed using semi-structured interviews assessing staff experience with workflow and adoption of Foundations of Fitness Program.
Fidelity to planned program | 24 weeks
  We will assess percent of planned class sessions and planned outcome assessments that were administered.

CONTACTS AND LOCATIONS:
Overall Officials: Auden C McClure, MD MPH, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No